CLINICAL TRIAL: NCT01531894
Title: An Open Label Continuation Study of the Oral AKT Inhibitor GSK2110183 in Subjects With Solid Tumors and Hematologic Malignancies
Brief Title: Continuation Study of the Oral AKT Inhibitor GSK2110183
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115131; 2014-002041-22 (EudraCT Number)
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: solid tumor; GSK2110183; hematologic malignancy; AKT inhibitor; cancer; safety
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — GSK2110183; afuresertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- GSK2110183 (afuresertib) (Experimental): All patients received the GSK2110183 (afuresertib) treatment
  Interventions: Drug: GSK2110183 (afuresertib)

INTERVENTIONS:
Drug: GSK2110183 (afuresertib) — Afuresertib is an oral, low nanomolar pan-AKT kinase inhibitor immediate release (IR) 50 mg or 75 mg tablets was to be taken orally with at least 200 mL of water, with or without food, in the morning.
  Other Names: ASB183

SUMMARY:
This multicenter, non-randomized, open-label, treatment continuation or 'rollover' study was designed to provide continued access to eligible subjects who had previously participated in a GSK2110183 study (parent study) sponsored by GlaxoSmithKline (GSK) or another research organization working on behalf of GSK. Eligible subjects had previously received clinical benefit from continued treatment and had to have ad an acceptable safety profile with GSK2110183. Subjects who had participated in a GSK2110183 combination study with an approved anti-cancer agent were also be eligible to enroll in this rollover study. Subjects who participated in combination studies with two investigational compounds (one being GSK2110183) were not eligible for this rollover study. Subjects were enrolled by cohort based on the duration and treatment received while in their parent study. Safety assessments (physical examinations, vital sign measurements, 12-lead electrocardiograms, echocardiograms or multiple-gated acquisition scans, clinical laboratory assessments and monitoring of adverse events) were evaluated during this study. Disease assessment were performed using local standard of care imaging practices and criteria appropriate for disease type and location.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed informed consent for this study.
* Is currently participating in a GSK2110183 study (monotherapy or in combination with an approved anti-cancer agent) sponsored by GSK or by another research organization working on behalf of GSK.
* Currently benefitting from continued treatment and have an acceptable safety profile with GSK2110183 as determined by the investigator following previous treatment with GSK2110183 either as monotherapy or as part of a combination treatment regimen.
* Continued ability to swallow and retain orally administered study treatment(s) and does not have any clinically significant GI abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Male subjects with a female partner of childbearing potential must be willing to continue practicing the same acceptable method of contraception as used in the parent study during the rollover study and for at least 16 weeks after the last dose of GSK2110183.
* Female subjects of childbearing potential, as defined in the parent study, must be willing to continue practicing the same acceptable method of contraception as used in the parent study during the rollover study and for at least 4 weeks after the last dose of GSK2110183.
* Female subjects of childbearing potential, as defined in parent study, must have negative serum pregnancy tests at the time of transition to this study.
* Maintain a performance status score of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) scale
* Subjects with Type II diabetes are only allowed if their HbA1C is less than 8 percent at study entry.
* Have adequate organ system function

Exclusion Criteria:

* Permanent discontinuation of GSK2110183 in the parent study due to toxicity or disease progression.
* Concomitant use of any type of anti-cancer treatment other than studied in the parent protocol.
* Local access to commercially available GSK2110183.
* Current use of a prohibitive medication(s)
* Current use of anticoagulants
* Any unresolved toxicity greater than Grade 2 , except for alopecia, (National Cancer Institute-Common Toxicity Criteria for Adverse Events [NCI-CTCAE], version 4.0) from parent study treatment at the time of transition to this study.
* History of HIV infection.
* Peripheral neuropathy greater than Grade 1
* History of hepatitis B or C infection (subjects with evidence of cleared hepatitis B are permitted).
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable, or uncompensated respiratory, hepatic, renal, metabolic or cardiac disease).
* QTcF interval greater than 500 msecs at the time of transition to this study.
* Other clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
* Evidence of current Class II, III, or IV heart failure as defined by the New York Heart Association [NYHA, 1994] functional classification system at the time of transition to this study.
* Symptomatic or untreated leptomeningeal, CNS or brain metastases or spinal cord compression at the time of transition to this study.
* Lactating female or female who becomes pregnant prior to transition to this study.
* Previously diagnosed diabetes mellitus Type I. Subjects with Type II diabetes are allowed if entry criteria are fulfilled
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions at the time of transition to this study that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator or GSK Medical Monitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02-08 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (3):
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Galway, Ireland
- Novartis Investigative Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As this was a rollover study, there was no planned number of subjects. Eleven subjects were enrolled and analyzed in the study.
Pre-assignment Details: There was no planned duration of treatment as this was a rollover study. The subjects could permanently discontinue the study treatment due to protocol deviation, adverse event, disease progression, withdrawal of consent, Investigator's discretion, lost to follow-up, termination of study or death.
Period: Overall Study
Arm/Group | GSK2110183 (Afuresertib)
Started | 11
Completed | 2
Not Completed | 9
Not completed — Physician Decision | 8
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The 'all treated subjects' population consisted of all subjects that received at least one dose of afuresertib in this rollover study.
Arm/Group | GSK2110183 (Afuresertib)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian heritage | 2
  White - White/Caucasian/European heritage | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Events (AEs)
Description: Adverse Events (AEs) includes Summary of adverse events, drug related AEs, Serious adverse events, adverse events leading to study treatment discontinuation and death.
Time Frame: from the time of consent until the final study visit up to approx. 76 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2110183 (Afuresertib)
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 2239 days.
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of about 76 months.
Groups:
- All Patients: All patients received the GSK2110183 (afuresertib) treatment
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=11)
Gastritis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=11)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal discomfort (Gastrointestinal disorders) | 1
Oesophageal pain (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 2
Fatigue (General disorders) | 5
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Peripheral swelling (General disorders) | 1
Chronic sinusitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Ageusia (Nervous system disorders) | 1
Anosmia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT01531894/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT01531894/SAP_001.pdf